CLINICAL TRIAL: NCT03640884
Title: Post-marketing Safety Surveillance of Xueshuantong-Injection : a Registry Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Xueshuantong--V2.0
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Adverse Drug Event; Adverse Drug Reactions; Anaphylactic Reaction; Severe Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Whole blood sample of the patient with severe adverse event
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xueshuantong-Injection: Patients who received the Xueshuantong-Injection for treatment will be consecutive included in this registry. The investigators will record all the information about ADR, application of Xueshuantong-Injection and the combined medications, etc.
  Interventions: Drug: Xueshuantong-Injection

INTERVENTIONS:
Drug: Xueshuantong-Injection — Xueshuantong-Injection is a kind of natural compound injection extracted from Chinese herb Notoginseng. The major bioactive ingredient is panax notoginseng saponins.
  Other Names: Chenzhong

SUMMARY:
This registry aims to monitor the safety of Xueshuantong Injection and to identify the potential risk factors for the adverse drug reactions.

DETAILED DESCRIPTION:
Xueshuantong-Injection is a kind of natural compound injection with Panax notoginseng saponins(PNS). It's a popular drug for improving blood circulation that focusing on central retinal vein occlusion, stroke sequela, internal ophthalmopathy, hyphema and so on. However, more and more case reports about the adverse drug events of Panax notoginseng saponins have been reported in recent years. Therefore, this registry of Xueshuantong-Injection aims to monitor the safety and find the incidence of adverse drug reactions to Xueshuantong-Injection. Moreover, this registry is highly concerned on identifying the potential risk factors for the adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use Xueshuantong-Injection in the monitoring departments of certain hospitals

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received the Xueshuantong-Injection for treatment will be consecutive included in this registry
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe adverse reactions (SAR) of Xueshuantong-Injection | 2 years
  A serious adverse reactions (SAR) is any untoward medical occurrence suspected to be medicinal product-related that at any dose: Results in death, is life-threatening, NOTE: The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. Requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or Is a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
The incidence of adverse drug reactions (ADR) of Xueshuantong-Injection | 2 years
The incidence of adverse events （AE）of Xueshuantong-Injection | 2 years
The incidence of serious adverse events （SAE）of Xueshuantong-Injection | 2 years
The incidence of anaphylactic reaction of Xueshuantong-Injection | 2 years
The incidence of new ADRs of Xueshuantong-Injection | 2 years
The effective rate of Xueshuantong-Injection | 2 years
  The proportion of the patients whose drug effect is considered as "effective" by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, M.D., Study Director — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Jinmin Liu, M.D., Principal Investigator — Dongfang Hospital Affiliated to Beijing University of traditional Chinese medicine
Locations (14):
- China (14):
  - Jizhou City Hospital, Hengshui, Hebei
  - Tongbai County People's Hospital, Nanyang, Henan
  - Lingbao 3th People's Hospital, Sanmenxia, Henan
  - People's Hospital of Dancheng County, Zhoukou, Henan
  - Dongxihu District People's Hospital, Wuhan, Hubei
  - Donghai Country People's Hospital, Lianyungang, Jiangsu
  - People's Hospital of Yichun City, Yichun, Jiangxi
  - Central Hospital of Wafangdian City, Dalian, Liaoning
  - Lingyuan City Central Hospital, Lingyuan, Liaoning
  - Chinse Medical Hospital of Yangxin County, Binzhou, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Yangcheng County People's Hospital, Jincheng, Shanxi
  - Lingshi Country People's Hospital, Jinzhong, Shanxi
  - Shanxi Yuanping First People's Hospital, Yuanping, Shanxi